CLINICAL TRIAL: NCT04079426
Title: Innate Immunity in Acute Respiratory Distress Syndrome: A Translational Approach to Limit Inflammasome-dependent Lung Inflammation by Tetracycline
Brief Title: Tetracycline to Limit the Innate Immune Response in Acute Respiratory Distress Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Dr. Christian Bode, Principal Investigator, University of Bonn
Other Study IDs: BOST-002
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Adult Respiratory Distress Syndrome; Pneumonia; Sepsis
Keywords: inflammasome; Caspase; NLRP3; Antibiotics; Tetracycline
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia; Sepsis | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sampling of Blood and bronchoalveolar lavage — Multiplex assays for pro- and anti-inflammatory markers and incubation of immune cells isolated from serum and bronchoalveolar lavage fluid of patients with ARDS.

SUMMARY:
The acute respiratory distress syndrome (ARDS) is a severe form of respiratory failure with a mortality rate of approximately 40%. Despite advances in its supportive treatment such as lung protective ventilation or restrictive fluid management, no effective pharmacotherapy exists to treat ARDS. Emerging preclinical data indicates that excessive activation of the inflammasome-Caspase 1 pathway plays a key role in the development of ARDS. Tetracycline has anti-inflammatory properties via inhibiting inflammasome-caspase-1 activation. Since not much is known about the activation of the inflammasome in clinical ARDS, the purpose of this study is i) to investigate the the inflammasome-caspase-1 activation in clinical ARDS and ii) inhibit the innate immune response of alveolar leucocytes obtained by tetracycline from patients with ARDS

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Informed consent of the patient
* Diagnosis of ARDS for < 48 h

Exclusion Criteria:

* Age < 18 years
* Missing informed consent
* Immune therapy
* Autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants admitted to the Intensive Care Unit of the University Hospital of Bonn with an initial diagnosis of ARDS
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Cytokine Levels in Serum and bronchoalveolar fluid | 1 week
  determined by multiplex Assay [pg/ml]
Activation Status of immune cells from blood and bronchoalveolar fluid | 1 week
  incubation of immune cells with tetracycline and Determination of cytokines by multiplex assay [pg/ml]
Alarmins in Serum and bronchoalveolar fluid | 1 week
  Determination by western blot, qPCR or flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peukert K, Fox M, Schulz S, Feuerborn C, Frede S, Putensen C, Wrigge H, Kummerer BM, David S, Seeliger B, Welte T, Latz E, Klinman D, Wilhelm C, Steinhagen F, Bode C. Inhibition of Caspase-1 with Tetracycline Ameliorates Acute Lung Injury. Am J Respir Crit Care Med. 2021 Jul 1;204(1):53-63. doi: 10.1164/rccm.202005-1916OC. PMID 33760701